CLINICAL TRIAL: NCT02171104
Title: MT2013-31: Allogeneic Hematopoietic Cell Transplantation for Inherited Metabolic Disorders and Severe Osteopetrosis Following Conditioning With Busulfan (Therapeutic Drug Monitoring), Fludarabine +/- ATG
Brief Title: MT2013-31: Allo HCT for Metabolic Disorders and Severe Osteopetrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013LS104
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Mucopolysaccharidosis Disorders; Hurler Syndrome; Hunter Syndrome; Maroteaux Lamy Syndrome; Sly Syndrome; Alpha-Mannosidosis; Fucosidosis; Aspartylglucosaminuria; Glycoprotein Metabolic Disorders; Sphingolipidoses; Recessive Leukodystrophies; Globoid Cell Leukodystrophy; Metachromatic Leukodystrophy; Niemann-Pick B; Niemann-Pick C Subtype 2; Sphingomyelin Deficiency; Peroxisomal Disorders; Adrenoleukodystrophy With Cerebral Involvement; Zellweger Syndrome; Neonatal Adrenoleukodystrophy; Infantile Refsum Disease; Acyl-CoA Oxidase Deficiency; D-Bifunctional Enzyme Deficiency; Multifunctional Enzyme Deficiency; Alpha-methylacyl-CoA Racmase Deficiency; Mitochondrial Neurogastrointestingal Encephalopathy; Severe Osteopetrosis; Hereditary Leukoencephalopathy With Axonal Spheroids (HDLS; CSF1R Mutation); Inherited Metabolic Disorders
Keywords: allogeneic hematopoietic cell transplantation; bone marrow transplantation; IMD; AMACRD; MNGIE; HDLS; OP; ALD
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; alpha-Mannosidosis; Fucosidosis; Aspartylglucosaminuria; Sphingolipidoses; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Peroxisomal Disorders; Zellweger Syndrome; Refsum Disease, Infantile; Peroxisomal ACYL-COA oxidase deficiency; Pseudo-Zellweger syndrome; Osteopetrosis; Hereditary Diffuse Leukoencephalopathy with Spheroids; Alpha-Methylacyl-CoA Racemase Deficiency | interventions — Stem Cell Transplantation; Regimen B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- IMD - Except Haplo-identical (Experimental): Inherited Metabolic Disease (IMD) - Except Haplo-Identical
  See intervention descriptions.
  Interventions: Biological: Stem Cell Transplantation; Drug: IMD Preparative Regimen
- OP - Except Haplo-Identical (Experimental): Severe Osteoperosis (OP) - Except Haplo-Identical
  See intervention descriptions.
  Interventions: Biological: Stem Cell Transplantation; Drug: Osteopetrosis Only Preparative Regimen
- OP and IMD -Haplo-Identical Only (Experimental): Severe Osteopetrosis (OP) and Inhterited Metabolic Disorders (IMD)
  -Haplo-Identical Only
  See intervention descriptions.
  Interventions: Biological: Stem Cell Transplantation; Drug: Osteopetrosis Haploidentical Only Preparative Regimen
- cALD SR-A (Standard-Risk, Regimen A) (Experimental): See intervention descriptions.
  Interventions: Biological: Stem Cell Transplantation; Drug: IMD Preparative Regimen; Drug: cALD SR-A (Standard-Risk, Regimen A)
- cALD SR-B (Standard-Risk, Regimen B) (Experimental): See intervention descriptions.
  Interventions: Biological: Stem Cell Transplantation; Drug: IMD Preparative Regimen; Drug: cALD SR-B (Standard-Risk, Regimen B)
- cALD HR-C (High-Risk, Regimen C) (Experimental): See intervention descriptions.
  Interventions: Biological: Stem Cell Transplantation; Drug: IMD Preparative Regimen; Drug: cALD HR-D (High-Risk, Regimen C)
- cALD HR-D (High-Risk, Regimen D) (Experimental): See intervention descriptions.
  Interventions: Biological: Stem Cell Transplantation; Drug: IMD Preparative Regimen; Drug: cALD HR-D (High-Risk, Regimen D)

INTERVENTIONS:
Biological: Stem Cell Transplantation — Infusion given on Day 0
Drug: IMD Preparative Regimen — * Anti-thymocyte Globulin (ATG)
  * Fludarabine
  * Busulfan
  Arms: IMD - Except Haplo-identical; cALD HR-C (High-Risk, Regimen C); cALD HR-D (High-Risk, Regimen D); cALD SR-A (Standard-Risk, Regimen A); cALD SR-B (Standard-Risk, Regimen B)
Drug: Osteopetrosis Only Preparative Regimen — * Anti-thymocyte Globulin (ATG)
  * Fludarabine
  * Busulfan
  * Thiotepa
  Arms: OP - Except Haplo-Identical
Drug: Osteopetrosis Haploidentical Only Preparative Regimen — * Rituximab
  * Alemtuzumab
  * Busulfan
  * Fludarabine
  Arms: OP and IMD -Haplo-Identical Only
Drug: cALD SR-A (Standard-Risk, Regimen A) — N-acetylcysteine start day +1 through day +28
  Arms: cALD SR-A (Standard-Risk, Regimen A)
Drug: cALD SR-B (Standard-Risk, Regimen B) — N-acetylcysteine start day +1through day +56
  Arms: cALD SR-B (Standard-Risk, Regimen B)
Drug: cALD HR-D (High-Risk, Regimen C) — N-acetylcysteine and celecoxib start day of admission (prior to conditioning regimen) and continue through day +100
  Arms: cALD HR-C (High-Risk, Regimen C)
Drug: cALD HR-D (High-Risk, Regimen D) — N-acetylcysteine, celecoxib, vitamin E and alpha lipoic acid start day of admission (prior to conditioning regimen) and continue through day +100
  Arms: cALD HR-D (High-Risk, Regimen D)

SUMMARY:
This single-institution, phase II study is designed to test the ability to achieve donor hematopoietic engraftment while maintaining low rates of transplant-related mortality (TRM) using busulfan- and fludarabine-based conditioning regimens with busulfan therapeutic drug monitoring (TDM) for patients with various inherited metabolic disorders (IMD) and severe osteopetrosis (OP).

ELIGIBILITY:
Inclusion Criteria:

* 0 through 55 years of age
* Adequate graft available
* Adequate organ function
* Eligible Diseases:

  * Mucopolysaccharidosis Disorders:

    * MPS IH (Hurler syndrome)
    * MPS II (Hunter syndrome) if the patient has no or minimal evidence of symptomatic neurologic disease but is expected to have a neurologic phenotype
    * MPS VI (Maroteaux-Lamy syndrome)
    * MPS VII (Sly syndrome)
  * Glycoprotein Metabolic Disorders:

    * Alpha mannosidosis
    * Fucosidosis
    * Aspartylglucosaminuria
  * Sphingolipidoses and Recessive Leukodystrophies:

    * Globoid cell leukodystrophy
    * Metachromatic leukodystrophy
    * Niemann-Pick B patients (sphingomyelin deficiency)
    * Niemann-Pick C subtype 2
  * Peroxisomal Disorders:

    * Adrenoleukodystrophy with cerebral involvement
    * Zellweger syndrome
    * Neonatal Adrenoleukodystrophy
    * Infantile Refsum disease
    * Acyl-CoA-Oxidase Deficiency
    * D-Bifunctional enzyme deficiency
    * Multifunctional enzyme deficiency
    * Alpha-methylacyl-CoA Racmase Deficiency (AMACRD)
    * Mitochondrial Neurogastrointestingal Encephalopathy (MNGIE)
  * Severe Osteopetrosis (OP)
  * Hereditary Leukoencephalopathy with axonal spheroids (HDLS; CSF1R mutation)
  * Other Inherited Metabolic Disorders (IMD): Patients will also be considered who have other life-threatening, rare lysosomal, peroxisomal or other similar inherited disorders characterized by white matter disease or other neurologic manifestations for which there is rationale that transplantation would be of benefit, such as certain patients with Wolman's disease, GM1 gangliosidosis, I-cell disease, Tay-Sachs disease, Sandhoff disease or others.
  * Voluntary written consent

Exclusion Criteria:

* Pregnancy - menstruating females must have a negative serum or urine pregnancy test within 14 days of study treatment start
* Prior myeloablative chemotherapy exposure within 4 months of the start of conditioning on this protocol (patients excluded for this reason may be eligible for other institutional protocols)
* Uncontrolled bacterial, fungal or viral infections including HIV (including active infection with Aspergillus or other mold within 30 days)

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 149 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2029-07-14 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects who achieve high-level donor hematopoietic engraftment | Day +42 post-transplant
  Defined as neutrophil recovery by Day +42 post-transplant and ≥ 80% donor cells on the myeloid fraction of peripheral blood at Day +100 post-transplant
Percent of subjects who achieve high-level donor hematopoietic engraftment | Day +100 post-transplant
  Defined as ≥ 80% donor cells on the myeloid fraction of peripheral blood at Day +100 post-transplant

SECONDARY OUTCOMES:
Graft-versus-host disease | Day +100 post-transplant
  Incidence and severity of GvHD
Transplant-related mortality | Day +100 post-transplant
  Incidence of TRM
Regimen-related toxicity | Day +100 post-transplant
  Defined as infection, acute renal failure, respiratory failure, cardiac failure, and veno-occlusive disease
Post-HSCT changes in disease | 1 year
  Incidence of radiographic, physiologic, neuro-psychologic, and/or biochemical aspects of the disease as assessed on a disease-specific basis
Post-HSCT changes in disease | 2 years
  Incidence of radiographic, physiologic, neuro-psychologic, and/or biochemical aspects of the disease as assessed on a disease-specific basis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States